CLINICAL TRIAL: NCT05343767
Title: A Phase II, Randomized, Double Blind, Double Dummy, Active-Controlled Clinical Trial to Investigate the Efficacy and Safety of Low-Glu in Patients Newly Diagnosed With Type II Diabetes Mellitus
Brief Title: Investigate the Efficacy and Safety of Low-Glu in Patients Newly Diagnosed With Type II Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Natural Wellness Egypt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NW_Low-Glu_14122016
Record Dates: First submitted 2022-04-10; First posted 2022-04-25 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Type2 Diabetes Mellitus
Keywords: Ficus deltoidea; HbA1c; weight; metabolic syndrome; medicinal plants
MeSH Terms: conditions — Body Weight; Metabolic Syndrome | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: This was a double-blind, double dummy, randomized, active-controlled, three-arm, parallel-group, interventional phase II clinical trial to investigate efficacy and safety of a herbal medicinal product of (NW Low-Glu) in patients newly diagnosed with type II diabetes mellitus.
  Study duration: 3 months of recruitment and 3 months of treatment. Sample Size: It was planned to enroll 68 patients per arm, 204 in total. Participants were patients between 18 and 65 years of age, newly diagnosed with type II diabetes mellitus and consenting to participate in this study.
  Eligible patients were randomized in a 1:1:1 allocation ratio, into one of the three treatment groups, to receive either Metformin or one of the two doses of NW Low-Glu.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization was done using interactive response technology (IWRS).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Arm 1 Metformin ( 64 patients) (Active Comparator): Metformin 1000 mg tablets were used.
  * First Dose: One Metformin 1000 mg tablet + Two Placebo Capsules administered PO on empty stomach with plenty of water 2 hours after meals.
  * Second Dose: Two Placebo Capsules administered PO on empty stomach with plenty of water 2 hours after meals.
  * Third Dose: One Metformin 1000 mg tablet + Two Placebo Capsules administered PO on empty stomach with plenty of water 2 hours after meals.
  A total dose of 2000 mg was administered per day.
  Interventions: Other: Metformin
- Experimental Arm 2: Low Dose NW Low-Glu ( 65 patients) (Experimental): The contents of 4 capsules of NW Low-Glu were equally distributed and inserted into 6 capsules size 0, and administered in 3 daily doses as follows:
  * First Dose: One Placebo tablet + Two size 0 NW Low-Glu Capsules administered PO on empty stomach with plenty of water 2 hours after meals.
  * Second Dose: Two size 0 NW Low-Glu Capsules administered PO on empty stomach with plenty of water 2 hours after meals.
  * Third Dose: One Placebo tablet + Two size 0 NW Low-Glu Capsules administered PO on empty stomach with plenty of water 2 hours after meals.
  Interventions: Dietary Supplement: Natural Wellness Low-Glu low dose
- Experimental Arm 3: High Dose NW Low-Glu ( 69 patients) (Experimental): The contents of 5 capsules of NW Low-Glu were equally distributed and inserted into 6 capsules size 0, and administered in 3 daily doses as follows:
  * First Dose: One Placebo tablet + Two size 0 NW Low-Glu Capsules administered PO on empty stomach with plenty of water 2 hours after meals.
  * Second Dose: Two size 0 NW Low-Glu Capsules administered PO on empty stomach with plenty of water 2 hours after meals.
  * Third Dose: One Placebo tablet + Two size 0 NW Low-Glu Capsules administered PO on empty stomach with plenty of water 2 hours after meals.
  Interventions: Dietary Supplement: Natural Wellness Low-Glu high dose

INTERVENTIONS:
Dietary Supplement: Natural Wellness Low-Glu low dose — The contents of 4 capsules of NW Low-Glu were equally distributed and inserted into 6 capsules size 0, and administered in 3 daily doses
  Other Names: Mas Cotek powdered Extract 300 mg + Cinnamomum cassia L. powdered Extract 100 mg + Black seed powdered extract 250 mg
  Arms: Experimental Arm 2: Low Dose NW Low-Glu ( 65 patients)
Dietary Supplement: Natural Wellness Low-Glu high dose — The contents of 5 capsules of NW Low-Glu were equally distributed and inserted into 6 capsules size 0, and administered in 3 daily doses
  Arms: Experimental Arm 3: High Dose NW Low-Glu ( 69 patients)
Other: Metformin — A total dose of 2000 mg was administered per day.
  Arms: Control Arm 1 Metformin ( 64 patients)

SUMMARY:
Ficus deltoidea leaves, Cinnamomum cassia and Black seed powdered extract have long been used for the treatment of type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Diabetes Mellitus (DM), commonly referred to as Diabetes is defined by World Health Organization (WHO) as a group of metabolic disorders characterized by chronic Hyperglycemia resulting from defects in insulin secretion, insulin action or both. Long-term organ damage, organ dysfunction and organ failure are associated with the chronic Hyperglycemia of Diabetes. Possible Diabetes complications can be classified into two major categories; macrovascular and microvascular including Ischemic Heart Disease (IHD), Peripheral Vascular Disease (PVD), and Cerebrovascular Disease (CVD) "macrovascular", and Nephropathy, Retinopathy, and Neuropathy "microvascular" resulting in organ and tissue damage in almost one third to one half of population with diabetes.

According to the International Diabetes Federation (IDF), the three main types of Diabetes are Type 1 Diabetes, Type 2 Diabetes and Gestational Diabetes. Type 1 DM, formerly described as "Insulin Dependent Diabetes Mellitus" (IDDM) results from β-cells destruction, usually leading to absolute deficiency of insulin. Type 2 DM formerly described as "Non-Insulin-Dependent Diabetes Mellitus" (NIDDM) results from a progressive insulin secretory defect on the background of insulin resistance. Gestational Diabetes, which appears during pregnancy, is associated with increasing the risk of developing type 2 Diabetes in both mother and child later in life.

Diabetes is a rapidly growing health concern in both developed and developing nations and its prevalence is continuously increasing worldwide. Globally, in 2014, approximately 422 million adults were having diabetes, with type 2 making up about 91%of the cases. In 2015, according to IDF, an estimated 415 million adults were having diabetes along with an estimated 318 million adults with impaired glucose tolerance. Both WHO and IDF predict that by 2030, this number will be doubled. In 2016 the WHO global report on Diabetes stated that the prevalence of Diabetes has increased faster in low- and middle-income countries than in high-income countries.

Type 2 Diabetes is characterized by insulin resistance and/or abnormal insulin secretion, either of which may predominate. It is associated with several metabolic defects such as obesity, hypertension, and dyslipidemia, which contribute to the very high rate of cardiovascular morbidity and mortality.

Medicinal herbs were used to treat a wide range of diseases long time before the birth of conventional medicine systems. The World Health Organization (WHO) has listed 21,000 plant names, which are used for medicinal purposes around the world, so despite the fact that medicinal herbs are at times misconceived as being unscientific, their continual existence proves they are able to be alternatives or complementary to conventional drugs at some point.

Specifically, Ficus deltoidea leaves, Cinnamomum cassia L. powdered Extract and Black seed powdered extract have been used for the treatment of Diabetes Mellitus and other medical conditions for over 2000 years. Ficus deltoidea is an evergreen shrub reaching to 2 meters of height, with whitish grey bark, broadly spoon-shaped to obovate leaves and spherical or round figs. Over the years, it has been used to treat many diseases such as; Diabetes Mellitus, Hypertension, Hyperlipidemia and Gout. Numerous studies were conducted over the past years to assess the safety of Ficus deltoidea, Cinnamomum cassia L. powdered extract and Black seed powdered extract and their efficacy in treating type 2 Diabetes Mellitus.

As the available data on NW Low-Glu efficacy, safety and dosing regimen is not enough, this study will be conducted to compare the hypoglycemic effect of two doses of a herbal medicinal product of ficus and Cinnamomum cassia L. powdered Extract + Black seed powdered extract (NW Low-Glu) to that of Metformin as measured by the mean change in HbA1c levels in patients newly diagnosed with type II diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent.
2. Males and females aged between 18 and 65 years of age.
3. Newly diagnosed with type II diabetes mellitus patients as per the following criteria (FBG ≥ 126 mg/dl) or, 2h- post prandial ≥ 200 mg/dl during OGTT or, HbA1c ≥ 6.5%
4. Anti-diabetic treatment naïve patients.
5. Able and willing to perform SMBG and to complete subject diaries.

Exclusion Criteria:

1. Pregnant or lactating women; women of childbearing potential must agree to use an accepted method of contraception during the course of the study and for 1 month after their last dose of study drug.
2. Patients with BMI > 40 Kg/m2 or BMI < 18.5 Kg/m2.
3. eGFR <60 mL/min/1.73 m2 (measured by the CKD-EPI equation) 3.
4. History of Positive human immunodeficiency virus, hepatitis B surface antigen (HBsAG), or hepatitis C antibody test.
5. History of type I diabetes, diabetes resulting from pancreatic injury, or secondary forms of diabetes such as Cushing's syndrome or acromegaly.
6. History of diabetic complications such as diabetic ketoacidosis, lactic acidosis or state of hyperosmolar hyperglycemia, diabetic proliferative retinopathy, or severe diabetic neuropathy (requiring treatment with antidepressants or opioids) and history of decompensated diabetes (polyuria, polydipsia, nocturia, fatigue).
7. History of chronic gastrointestinal (GI) conditions that could impede gastric emptying or potentially affect the interpretation of the study data.
8. History of weight loss surgery or weight loss procedure involving the GI tract, such as gastric bypass, gastric stapling, or gastric banding.
9. History of an eating disorder (e.g., bulimia, anorexia).
10. History of malignancy (except treated basal or squamous cell skin cancer) within 5 years prior to screening.
11. History of significant cardiovascular disease (such as congestive heart failure, myocardial infarction, coronary disease) or uncontrolled hypertension.
12. History of clinically significant renal or liver disease.
13. Receipt of an investigational drug within 30 days prior to screening, or active enrollment in another investigational medication or device trial.
14. Known or suspected allergy to the trial products.
15. Any condition, in the judgment of the investigator, that would interfere with the patient's ability to comply with all study requirements or that would place the patient at unacceptable risk by his/her participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
To compare the hypoglycemic effect of two doses of a herbal medicinal product (NW Low-Glu) to that of Metformin as measured by the mean change in HbA1c levels in patients newly diagnosed with type II diabetes mellitus. | 12 weeks
  Comparing the mean change in HbA1c levels between each experimental arm and active-control arm

SECONDARY OUTCOMES:
To measure the incidence of hypoglycemia events and other adverse events in patients newly diagnosed with type II diabetes mellitus (Safety) | 12 weeks
  Comparing the mean change in fasting plasma glucose levels between each experimental arm and active-control arm
To compare the mean change in the 2h-post prandial glucose levels between each experimental arm and active-control arm (efficacy) | 12 weeks
  To compare the mean change in the 2h-post prandial glucose levels between each experimental arm and active-control arm.

OTHER OUTCOMES:
Exploratory outcome | 12 weeks
  To explore the effect of NW Low-Glu on Beta cell function in patients newly diagnosed with type II diabetes mellitus by assessing through HOMA-β modeling.
Measuring the activity of alpha-glucosidase enzyme to investigate the effect of NW Low-Glu on intestinal glucose absorption | 12 weeks
  To investigate the effect of NW Low-Glu on intestinal glucose absorption by measuring the activity of alpha-glucosidase enzyme.
To investigate the effect of NW Low-Glu on weight. | 12 weeks
  To investigate the effect of NW Low-Glu on weight by comparing patients' weight before and after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr Samir Helmy Assaad, MD, Principal Investigator — University of Alexandria
Locations (1):
- Natural Welness Egypt, Cairo, Nasr City, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cade WT. Diabetes-related microvascular and macrovascular diseases in the physical therapy setting. Phys Ther. 2008 Nov;88(11):1322-35. doi: 10.2522/ptj.20080008. Epub 2008 Sep 18. PMID 18801863
- [Background] Alberti KG, Zimmet PZ. Definition, diagnosis and classification of diabetes mellitus and its complications. Part 1: diagnosis and classification of diabetes mellitus provisional report of a WHO consultation. Diabet Med. 1998 Jul;15(7):539-53. doi: 10.1002/(SICI)1096-9136(199807)15:73.0.CO;2-S. PMID 9686693
- [Background] IDF. IDF Diabetes Atlas · Seventh Edition. 2015.
- [Background] WHO. Global report on diabetes. 2016.
- [Background] Shaw JE, Sicree RA, Zimmet PZ. Global estimates of the prevalence of diabetes for 2010 and 2030. Diabetes Res Clin Pract. 2010 Jan;87(1):4-14. doi: 10.1016/j.diabres.2009.10.007. Epub 2009 Nov 6. PMID 19896746
- [Background] Zimmet P, Alberti KG, Shaw J. Global and societal implications of the diabetes epidemic. Nature. 2001 Dec 13;414(6865):782-7. doi: 10.1038/414782a. PMID 11742409
- [Background] Edelman SV. Type II diabetes mellitus. Adv Intern Med. 1998;43:449-500. PMID 9506190
- [Background] Pan SY, Pan S, Yu ZL, Ma DL, Chen SB, Fong WF, Han YF, Ko KM. New perspectives on innovative drug discovery: an overview. J Pharm Pharm Sci. 2010;13(3):450-71. doi: 10.18433/j39w2g. PMID 21092716
- [Background] Bamosa A, Kaatabi H, Badar A, Al-Khadra A, Al Elq A, Abou-Hozaifa B, Lebda F, Al-Almaie S. Nigella sativa: A potential natural protective agent against cardiac dysfunction in patients with type 2 diabetes mellitus. J Family Community Med. 2015 May-Aug;22(2):88-95. doi: 10.4103/2230-8229.155380. PMID 25983604
- [Background] Jia Q, Liu X, Wu X, Wang R, Hu X, Li Y, Huang C. Hypoglycemic activity of a polyphenolic oligomer-rich extract of Cinnamomum parthenoxylon bark in normal and streptozotocin-induced diabetic rats. Phytomedicine. 2009 Aug;16(8):744-50. doi: 10.1016/j.phymed.2008.12.012. Epub 2009 May 22. PMID 19464860
- [Background] Corner E. The complex of Fixcus Deltoidea ; A recent invasion of the sunda shelf. Philos Trans R Soc London B, Biol Sci. 1969 Nov;256(808):281-317.
- [Background] Hakiman M, Maziah M. Non enzymatic and enzymatic antioxidant activities in aqueous extract of different Ficus deltoidea accessions. J Med Plants Res. 2009;3(3):120-31.
- [Background] Sulaiman MR, Hussain MK, Zakaria ZA, Somchit MN, Moin S, Mohamad AS, Israf DA. Evaluation of the antinociceptive activity of Ficus deltoidea aqueous extract. Fitoterapia. 2008 Dec;79(7-8):557-61. doi: 10.1016/j.fitote.2008.06.005. Epub 2008 Jul 10. PMID 18672036
- [Background] Prakash B, Singh P, Yadav S, Singh SC, Dubey NK. Safety profile assessment and efficacy of chemically characterized Cinnamomum glaucescens essential oil against storage fungi, insect, aflatoxin secretion and as antioxidant. Food Chem Toxicol. 2013 Mar;53:160-7. doi: 10.1016/j.fct.2012.11.044. Epub 2012 Dec 5. PMID 23220615
- [Background] Tauseef Sultan M, Butt MS, Anjum FM. Safety assessment of black cumin fixed and essential oil in normal Sprague Dawley rats: Serological and hematological indices. Food Chem Toxicol. 2009 Nov;47(11):2768-75. doi: 10.1016/j.fct.2009.08.011. Epub 2009 Aug 21. PMID 19699773
- [Background] Draman S, Aris M, Razman, SFU A, H A, AR NA, et al. Mas Cotek (Ficus deltoidea): A Possible Supplement for Type II Diabetes: (A Pilot Study). Pertanika J Trop Agric Sci. 2012;35(1):93-102.
- [Background] Monnier L, Colette C. Target for glycemic control: concentrating on glucose. Diabetes Care. 2009 Nov;32 Suppl 2(Suppl 2):S199-204. doi: 10.2337/dc09-S310. No abstract available. PMID 19875552
- [Background] American Diabetes Association. 9. Pharmacologic Approaches to Glycemic Treatment: Standards of Medical Care in Diabetes-2021. Diabetes Care. 2021 Jan;44(Suppl 1):S111-S124. doi: 10.2337/dc21-S009. PMID 33298420
- [Background] Handelsman Y, Bloomgarden ZT, Grunberger G, Umpierrez G, Zimmerman RS, Bailey TS, Blonde L, Bray GA, Cohen AJ, Dagogo-Jack S, Davidson JA, Einhorn D, Ganda OP, Garber AJ, Garvey WT, Henry RR, Hirsch IB, Horton ES, Hurley DL, Jellinger PS, Jovanovic L, Lebovitz HE, LeRoith D, Levy P, McGill JB, Mechanick JI, Mestman JH, Moghissi ES, Orzeck EA, Pessah-Pollack R, Rosenblit PD, Vinik AI, Wyne K, Zangeneh F. AMERICAN ASSOCIATION OF CLINICAL ENDOCRINOLOGISTS AND AMERICAN COLLEGE OF ENDOCRINOLOGY--CLINICAL PRACTICE GUIDELINES FOR DEVELOPING A DIABETES MELLITUS COMPREHENSIVE CARE PLAN--2015--EXECUTIVE SUMMARY. Endocr Pract. 2015 Apr;21(4):413-37. No abstract available. PMID 27408942
- [Background] Bunawan H, Amin NM, Bunawan SN, Baharum SN, Mohd Noor N. Ficus deltoidea Jack: A Review on Its Phytochemical and Pharmacological Importance. Evid Based Complement Alternat Med. 2014;2014:902734. doi: 10.1155/2014/902734. Epub 2014 Mar 18. PMID 24772185
- [Background] Choo CY, Sulong NY, Man F, Wong TW. Vitexin and isovitexin from the Leaves of Ficus deltoidea with in-vivo alpha-glucosidase inhibition. J Ethnopharmacol. 2012 Aug 1;142(3):776-81. doi: 10.1016/j.jep.2012.05.062. Epub 2012 Jun 7. PMID 22683902
- [Background] Adam Z, Khamis S, Ismail A, Hamid M. Ficus deltoidea: A Potential Alternative Medicine for Diabetes Mellitus. Evid Based Complement Alternat Med. 2012;2012:632763. doi: 10.1155/2012/632763. Epub 2012 Jun 3. PMID 22701507
- [Background] Dugoua JJ, Seely D, Perri D, Cooley K, Forelli T, Mills E, Koren G. From type 2 diabetes to antioxidant activity: a systematic review of the safety and efficacy of common and cassia cinnamon bark. Can J Physiol Pharmacol. 2007 Sep;85(9):837-47. doi: 10.1139/Y07-080. PMID 18066129
- [Background] Crawford P. Effectiveness of cinnamon for lowering hemoglobin A1C in patients with type 2 diabetes: a randomized, controlled trial. J Am Board Fam Med. 2009 Sep-Oct;22(5):507-12. doi: 10.3122/jabfm.2009.05.080093. PMID 19734396
- [Background] Akilen R, Tsiami A, Devendra D, Robinson N. Cinnamon in glycaemic control: Systematic review and meta analysis. Clin Nutr. 2012 Oct;31(5):609-15. doi: 10.1016/j.clnu.2012.04.003. Epub 2012 May 12. PMID 22579946
- [Background] Askari G, Rouhani MH, Ghaedi E, Ghavami A, Nouri M, Mohammadi H. Effect of Nigella sativa (black seed) supplementation on glycemic control: A systematic review and meta-analysis of clinical trials. Phytother Res. 2019 May;33(5):1341-1352. doi: 10.1002/ptr.6337. Epub 2019 Mar 14. PMID 30873688
- [Background] Daryabeygi-Khotbehsara R, Golzarand M, Ghaffari MP, Djafarian K. Nigella sativa improves glucose homeostasis and serum lipids in type 2 diabetes: A systematic review and meta-analysis. Complement Ther Med. 2017 Dec;35:6-13. doi: 10.1016/j.ctim.2017.08.016. Epub 2017 Aug 30. PMID 29154069